CLINICAL TRIAL: NCT04532827
Title: The Effectiveness of Web-based Rehabilitation for Enhancing Workability and Daily Functioning for Persistent Physical Symptoms.
Brief Title: Web-based Rehabilitation for Persistent Physical Symptoms.
Acronym: DigiPimo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Finnish Institute of Occupational Health (Other)
Collaborators: The Social Insurance Institution of Finland (Unknown); the Hospital District of Helsinki and Uusimaa (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3531101
Record Dates: First submitted 2020-08-18; First posted 2020-08-31 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Persistent Physical Symptoms; Indoor Environment Associated Symptoms; Indoor Air Associated Symptoms; Chronic Fatigue Syndrome
Keywords: Indoor air; Persistent physical symptoms; Chronic Fatigue Syndrome; Web-based intervention; Rehabilitation; Indoor environment; EHealth
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The randomization will be pre-programmed and the allocation sequence will be carried out and concealed by a researcher who is not otherwise involved in trial at FIOH. This study compares eHealth intervention with treatment as usual. Thus it is not possible to blind the study participants. However, eHealth therapists are blinded for study participant compared with patients in eHealth intervention for other reasons, I.e. study participants and patients referred to the program as treatment as usual by their physician. Further, data analyst will be blinded to intervention arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case formulation with web-program (Experimental): The intervention will start with two video meetings with a psychologist to build up and present an individual case formulation, based on behavioural analysis, and to build up a shared decision of individual goals for the web program. The intervention continues with a web program consisting of ten manualized web-based modules, each at one-week intervals based on relational frame theory (RFT) and acceptance and commitment therapy (ACT). The pilot programme included six two-weeks modules and it was in use until 5/2021. The programme is in Finnish.
  Both participants in the intervention arm and in the treatment as the usual arm will receive usual care, meaning that TAU will be enhanced with the study intervention in the intervention arm. In addition to TAU, all participants will be given self-help and educational leaflet based on scientific knowledge related to their condition.
  Interventions: Behavioral: Case formulation with web-program
- Treatment as usual (No Intervention): Treatment as usual includes all the routine care that individual receives when he or she is presenting his or her symptoms at the primary or the occupational health care unit (corresponds primary care level treatment) or other unit that recommends the study for the participant. In practice, TAU may vary between the study participants based on their individual needs e.g. treatments for co-morbid somatic diseases or psychiatric disorders that this study will not interfere.
  Both participants in the intervention arm and in the treatment as usual arm will receive usual care, meaning that TAU will be enhanced with the study intervention in the intervention arm. In addition to TAU all participants will be given self-help and educational leaflet based on scientific knowledge related to their condition.

INTERVENTIONS:
Behavioral: Case formulation with web-program — The first meeting includes an interview to establish understanding on the participant´s symptomatology and current life situation, a case formulation (CF) will be build based on it. The CF is presented in the second session and modifications can be made to ensure acceptability for the participant. Goals for web program (WB) are set based on the CF and understanding of the factors contributing to the participant´s wellbeing.
  WB modules are instructed to complete during the week. Modules include psychoeducation, experiential exercises and training aimed at improving wellbeing and psychological flexibility. Web-therapist will offer written feedback. The participants can contact the therapist via the WB and al messages will be replied within one week. Automatic reminders will be sent if a participant has not been active in the WB, the therapists will call participants who have discontinued using the WB.
  Arms: Case formulation with web-program

SUMMARY:
Persistent physical symptoms (PPS) might diminish studying or workability and daily functioning without a clear medical or environment-related explanation. Psychosocial, patient-involving treatments that support individuals' abilities managing with the PPS and health behaviours have shown promising effects in treating PPS but the acceptability of these treatments among symptomatic individuals is low.

This study aims to assess the effectiveness of an eHealth intervention based on relational frame theory and acceptance and commitment therapy on PPS with two focus groups, among participants with indoor air associated disabling symptoms or persistent, chronic fatigue.

This study will compare web program enhanced with video-based individual case formulation with treatment as usual. The web program includes 10 one weeks (pilot included 6 two weeks) modules. In addition to patient-reported outcomes, ecological momentary assessments are conducted to provide real-time data on functioning and national registers are used to obtain information on health-care use and social benefits.

Data collection begins in August 2020 and will continue until 2023.

DETAILED DESCRIPTION:
Background: Frequent physical symptoms are common in the general population with over 90 per cent of the population reporting symptoms at some level. In some cases, they become persistent diminishing workability and daily functioning and associate with increased healthcare usage and sick leaves independently of other somatic or psychiatric comorbidities. Persistent physical symptoms (PPS) challenge health care systems as it is estimated that up to 4-30 per cent of primary health care visits are due to PPS without a clear medical explanation. Psychosocial, patient-involving treatments, such as cognitive-behavioural psychotherapy (CBT), that support individuals' abilities managing with the PPS and health behaviours have shown promising effects in treating PPS but so far, evidence-based treatments have resulted only in small to moderate effect sizes. The acceptability of these treatments among symptomatic individuals is also low - presumably because of the stigma related to the ambiguity of the PPS´ status as a medical condition. A stronger orientation to personalized treatment protocols is needed to improve the treatment efficacy and applicability.

This study will assess the effects of an eHealth intervention based on relational frame theory and acceptance and commitment therapy on PPS with two focus groups, among participants with indoor air associated disabling symptoms or persistent, chronic fatigue.

Methods: Using a randomized controlled design (RCT) with two parallel groups in a 1:1 ratio, the investigators will compare ACT/RFT-based web program enhanced with individual case formulation with treatment as usual. The web program intervention includes 10 one weeks (pilot included 6 two weeks) modules that each ask to complete the module and included training in two weeks. The web program is in Finnish. Participants will be asked to complete outcome questionnaires at baseline before the interview for inclusion, after the interview (randomization) and at 3, 6- and 12-months' follow-up after the randomization. The intervention group receives also a questionnaire four weeks after the beginning of the web program. In addition, ecological momentary assessments are also conducted to provide real-time data on functioning and national registers are used to obtain information on healthcare use and social benefits to complete patient-reported outcomes.

Eligible participants will be randomized to either the intervention or to TAU. The primary outcome will be a health-related quality of life. The secondary outcome measures are symptoms, illness perceptions, psychological flexibility and workability. Further, the investigators will assess whether any effect of the intervention on the primary outcome is mediated by the case formulation. The baseline data collection begins in August 2020 and will continue until 2022, follow-up data collection will continue until 2023.

ELIGIBILITY:
Inclusion Criteria:

* Fluent Finnish (web-program is in Finnish)
* Duration of the symptoms Onset of symptoms with disability maximum of 3 years before the study
* Symptomatology A) Indoor air-related symptoms or B) Persistent, chronic fatigue

A) Indoor air-related symptoms

1. Self-reported symptoms attributed to indoor (non-industrial) environments include: i) symptoms from at least two different organ systems eg. respiratory, digestive or nervous system.
2. Symptoms recurrently i) occur in more than one indoor environment or ii) continue despite environmental improvements (e.g. study or work arrangements and/or workplace repairs)

or

B) Chronic fatigue

1. Post-exertional malaise and/ or post-exertional fatigue.
2. Unrefreshing sleep or disturbance of sleep quantity or rhythm disturbance.
3. Multiorgan symptoms i) Pain, often widespread, ii) Two of more neurological or cognitive symptoms, iii) At least two symptoms of following categories: Autonomic manifestations, neuroendocrine manifestations or immune manifestations

   * Duration and severity of the condition: Symptoms minimum of six months; Symptoms are not lifelong and result in substantial functional restrictions in daily life.

Exclusion Criteria:

* Work situation: Long sick leave (≥3 months) without return to work plan, not actively participating in study or work life (retired or unemployed)
* Medical reasons

  1. Some serious and/or acute medical disease or illness explains the symptoms i) Somatic disease that explains the symptoms (e.g. uncontrolled asthma, hypothyroidism, sleep apnea)
  2. Psychiatric disorder (bipolar disorder, psychotic disorders, alcohol and/or drug dependency or abuse, eating disorders, and/or severe mood disorders)
  3. Developmental disorders
* Current psychotherapy
* Other Patient refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
The 15D questionnaire (health related quality of life) | Chance from baseline (i.e. at self-referral) to after randomisation (i.e. after clinical assessment), and to 6 and 14 weeks and to 6 and to 12 months after randomisation
  The 15D is a utility-based generic, standardized measure, comprising the following 15 dimensions that describe physical, mental, and social well-being: mobility, vision, hearing, breathing, sleeping, eating, speech, excretion, usual activities, mental function, discomfort and symptoms, depression, distress, vitality, and sexual activity. Each dimension is graded by the respondent on a scale ranging between 1 and 5, where 1 indicates an experience of no problems at all with the dimension and 5 indicates severe problems. Thus, the 15D can be used to measure a vast number of health states. We will use the 15D data both to derive 15D overall scores with values from 1 (full health) to 0 (being dead), and to obtain dimensional symptom profiles.

SECONDARY OUTCOMES:
Demographic questions: age (years) | At baseline (i.e. at self-referral)
Demographic questions: gender (male, female, prefer not to say) | At baseline (i.e. at self-referral)
Demographic questions: marital status (Unmarried, married or cohabiting, divorced or separation, widow) | At baseline (i.e. at self-referral)
Demographic questions: education (basic, secondary, higher) | At baseline (i.e. at self-referral)
Demographic questions: daily exercise | At baseline (i.e. at self-referral)
  One item of the frequency of the exercise on a six point likert scale (No weekly exercise - 4 times/week or more)
Demographic questions: Diet | At baseline (i.e. at self-referral)
  Two items of the diet on a six point likert scale (have daily regular eating habits - have no regular eating habits; Caffeine consumption never - 7 or more proportion per day)
Social support and loneliness | At baseline (i.e. at self-referral), and 12 months after randomisation
  Five questions of frequency of perceived loneliness and and social support in challenging situations (likert scale).
Smoking, Alcohol Use Disorders Identification Test (Audit-C) | At baseline (i.e. at self-referral), and 12 months after randomisation
Questions about health: Self-reported health | At baseline (i.e. at self-referral), and 12 months after randomisation
  Five point likert scale (very poor - very good)
Questions about health: Self-reported diseases (diagnosed by medical doctor) | At baseline (i.e. at self-referral), and 12 months after randomisation
Questions about health: medication | At baseline (i.e. at self-referral), and 12 months after randomisation
  Self-reported medication during past four weeks (name, dose, purpose of use)
Questions about health: Health care unit | At baseline (i.e. at self-referral), and 12 months after randomisation
  An open question of the participant´s health care provider.
Questions about health: Information seeking | At baseline (i.e. at self-referral), and 12 months after randomisation
  Questions about health information seeking from different sources (on a six point likert scale)
Questions about health: height in meters | At baseline (i.e. at self-referral)
  height in meters to calculate BMI kg/m^2
Questions about health: weight in kilograms | At baseline (i.e. at self-referral)
  weight in kilograms to calculate BMI kg/m^2
Work characteristics | At baseline (i.e. at self-referral), and 12 months after randomisation
  Questions about participant work characteristics (working hours, field of industry etc)
Symptoms related to environmental factors | At baseline (i.e. at self-referral), and 6 and 14 weeks and 6 and 12 months after randomisation
  Questions whether environmental factors such as mold or water damage in buildings, electromagnetic fields, chemicals or indoor air have associated with symptoms and have they associated with avoidance behavior (yes - no).
Health worries and health worries related to environmental factors | At baseline (i.e. at self-referral), and 14 weeks, and 6 and 12 months after randomisation
  Questions about health worries in general and related to environmental factors (scale 0 not worried at all - 10 extremely worried)
Environmental factors: influence on everyday life | At baseline (i.e. at self-referral), and 14 weeks, and 6 and 12 months after randomisation
  Questions about the influence of environmental factors on everyday life (scale 0 no consequences - 10 severe consequences)
Resiliency (SOC-3) | Time Frame: At baseline (i.e. at self-referral)
Personality Inventory (PK5) | Time Frame: At baseline (i.e. at self-referral)
Questions about sleep quality, sleeping patterns | At baseline (i.e. at self-referral), and 14 weeks, and, 6 and 12 months after randomisation
  Length of sleep (weekdays and weekends, hours)
Questions about sleep quality, sleeping patterns | At baseline (i.e. at self-referral), and 14 weeks, and 6 and 12 months after randomisation
  Nap (frequency per week and length, hours)
Questions about sleep quality, sleeping patterns | At baseline (i.e. at self-referral), and 14 weeks, and 6 and 12 months after randomisation
  Self-reported i) sleep quality, ii) night awakening iii) sleep disorders and iv) frequency of sleeping medicine usage at five point likert scale.
Questions about sleep quality, sleeping patterns | At baseline (i.e. at self-referral), and 14 weeks, and 6 and 12 months after randomisation
  Self-reported quality of rest and rhythmicity at four point likert scale.
Fatigue | At baseline (i.e. at self-referral), and 14 weeks, and 6 and 12 months after randomisation
  Questionnaire about perceived fatigue and its´consequences on daily functioning during past six months.
Generalized Anxiety Disorder 7 (GAD-7) | At baseline (i.e. at self-referral), and 14 weeks, and 6 and 12 months after randomisation
Insomnia Severity Index (ISI) | At baseline (i.e. at self-referral), and 14 weeks, and 6 and 12 months after randomisation
Patient Health Questionnaire-15 (PHQ-15) | At baseline (i.e. at self-referral), and 14 weeks, and 6 and 12 months after randomisation
The Patient Health Questionnaire (PHQ-9) | At baseline (i.e. at self-referral), and 14 weeks, and 6 and 12 months after randomisation
AIDO Healthcare app: daily mood and fatigue | 1.5, 3.5 and 12 months after randomisation
The Acceptance and Action Questionnaire -II AAQ-7 | At baseline (i.e. at self-referral), and 6 and 14 weeks and, 6 and 12 months after randomisation
Comprehensive assessment of Acceptance and Commitment Therapy CompACT | At baseline (i.e. at self-referral), and 14 weeks, 6 and 12 months after randomisation
Cognitive Fusion Questionnaire (CFQ-7) | At baseline (i.e. at self-referral), and 6 and 14 weeks and, 6 and 12 months after randomisation
Whiteley index -7 questionnaire | At baseline (i.e. at self-referral), and 14 weeks and 6 and 12 months after randomisation
White Bear Suppression Inventory (WBSI) | At baseline (i.e. at self-referral), after randomization and 14 weeks and, 6 and 12 months after randomisation
Five Facet Mindfulness Questionnaire (FFMQ) | At baseline (i.e. at self-referral), after randomization and 12 months after randomisation
Toronto alexithymia scale (TAS-20) | At baseline (i.e. at self-referral)
Illness Perception Questionnaire | At baseline (i.e. at self-referral) and 6 and 14 weeks and 6 and 12 months after randomisation
Self-assessed current ability to study or work | At baseline (i.e. at self-referral) and 14 weeks 6 and 12 months after randomisation
  One question about current ability to study or work on a scale 1-10.
Own prognosis of ability to study or work two years from now | At baseline (i.e. at self-referral) and 14 weeks 6 and 12 months after randomisation
  One question about of work ability two years from now (scale Unlikely; Not certain; Relatively certain)
Self-assessed stress and recovery | At baseline (i.e. at self-referral) and 14 weeks and 6 and 12 months after randomisation
  One question about stress and recovery on a scale 1-10.
Daily functioning in three sub-domains. | At baseline (i.e. at self-referral and 14 weeks and 6 and 12 months after randomisation
  Three questions about daily functioning (work, social life, home) on a scale 1-10 each
Working Alliance Inventory (WAI) - patient version for eHealth intervention | after randomization and 6 and 14 weeks after randomisation
Treatment satisfaction | after randomization and 6 and 14 weeks after randomisation
  Six items of treatment satisfaction based on Seligman´s report (1995). The effectiveness of psychotherapy: The Consumer Reports study. American psychologist, 50(12), 965.

OTHER OUTCOMES:
Interview of treatment acceptance | 12 months randomisation
  Interview for sample of intervention participants about the treatment acceptance (qualitative)
Engagement to the intervention | 14 weeks after randomisation.
  Total number of logins and time during the web-program, modules and exercises completed.
Reasons for discontinuing | Through study completion, an average of 1 year
  If participant discontinues he / she will be contacted.
The Finnish national health registers | At baseline (i.e. at self-referral), at 12 months after randomisation
  The Finnish national health registers to assess health care expenditures: Data on outpatient visits (AvoHILMO data), data on inpatient care (HILMO data), data on occupational health care use, information on prescribed and reimbursed prescription medicines purchases, information on rights for special reimbursement for medicines and information on sickness and disability benefits and rehabilitation with diagnoses

CONTACTS AND LOCATIONS:
Overall Officials: Tiina Paunio, Professor, Principal Investigator — University of Helsinki, Finnish Institute of Occupational Health, the Hospital District of Helsinki and Uusimaa
Locations (1):
- Finnish Institute of Occupational Health, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No
All IPD that underlie results in a publication could be published But: study participants choose in informed consent that do they accept that their IPD will be published (anonymized). If they choose 'no´, their data won´t be published. Thus the preliminary plan is not to share the IPD (´undecided' would be accurate as well).

REFERENCES:
- [Derived] Selinheimo S, Vuokko A, Lappalainen P, Keinonen K, Sainio M, Lappalainen R, Paunio T. The association between quality of life and psychological flexibility, depressive, anxiety or insomnia symptoms in patients with persistent indoor environment-related symptoms or chronic fatigue. BMC Psychol. 2025 Mar 11;13(1):229. doi: 10.1186/s40359-025-02549-8. PMID 40069901
- [Derived] Lappalainen P, Keinonen K, Lappalainen R, Selinheimo S, Vuokko A, Sainio M, Liesto S, Tolvanen A, Paunio T. Online acceptance and commitment therapy (iACT) for adults with persistent physical symptoms - 3-month follow-up study of a randomized controlled trial. J Psychosom Res. 2024 Aug;183:111830. doi: 10.1016/j.jpsychores.2024.111830. Epub 2024 Jun 13. PMID 38878337
- [Derived] Selinheimo S, Keinonen K, Vuokko A, Liesto S, Sainio M, Lappalainen R, Paunio T. A randomized controlled trial protocol for persistent physical symptoms associated with indoor environment or chronic fatigue: Effectiveness of video-based functional case conceptualization and web-program for improving quality of life. Front Psychol. 2023 Jan 6;13:923532. doi: 10.3389/fpsyg.2022.923532. eCollection 2022. PMID 36687807